CLINICAL TRIAL: NCT02845674
Title: An Open-Label Extension of a Randomized, Multicenter, Double-Masked, Vehicle-Controlled Study of the Safety and Efficacy of OTX-101 in the Treatment of Keratoconjunctivitis Sicca
Brief Title: An Open-Label Extension of a Phase 3 Study of OTX-101 in the Treatment of Keratoconjunctivitis Sicca
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTX-101-2016-002
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Keratoconjunctivitis Sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OTX-101 0.09% (Experimental): 0.09% cyclosporine nanomicellar solution
  Interventions: Drug: OTX-101 0.09%

INTERVENTIONS:
Drug: OTX-101 0.09% — 0.09% cyclosporine nanomicellar solution
  Other Names: Seciera

SUMMARY:
This is a safety extension enrolling subjects participating in Study OTX-101-2016-001 (NCT02688556)

ELIGIBILITY:
Inclusion Criteria:

* Completion of Study OTX-101-2016-001

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sheppard J, Bergmann M, Schechter BA, Luchs J, Ogundele A, Karpecki P. Phase 3 Efficacy (Worse-Eye Analysis) and Long-Term Safety Evaluation of OTX-101 in Patients with Keratoconjunctivitis Sicca. Clin Ophthalmol. 2021 Jan 12;15:129-140. doi: 10.2147/OPTH.S279364. eCollection 2021. PMID 33469259

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Group 1 and Group 2 consisted of subsets of subjects who received masked treatment with OTX-101 0.09% or with Vehicle, respectively, in OTX-101-2016-001. All subjects received open-label treatment with OTX-101 0.09% in OTX-101-2016-002.
Groups:
- OTX-101 0.09% to OTX-101 0.09%; Vehicle to OTX-101 0.09%: One drop in each eye BID
Period: Overall Study
Arm/Group | OTX-101 0.09% to OTX-101 0.09% | Vehicle to OTX-101 0.09%
Started | 129 | 129
Completed | 111 | 79
Not Completed | 18 | 50

BASELINE CHARACTERISTICS:
Population: Intent to treat population; Group 1 and Group 2 consisted of subsets of subjects who received masked treatment with OTX-101 0.09% or with Vehicle, respectively, in OTX-101-2016-001. All subjects received open-label treatment with OTX-101 0.09% in OTX-101-2016-002
Groups:
- Group 1: 0.09% cyclosporine nanomicellar solution
  OTX-101 0.09%: 0.09% cyclosporine nanomicellar solution
- Group 2: OTX-101 0.09%: 0.09% cyclosporine nanomicellar solution
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (15.51) | 61.5 (14.21) | 60.0 (14.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 107 | 216
  Male | 20 | 22 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 8 | 26
  Not Hispanic or Latino | 111 | 121 | 232
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 13 | 25
  White | 111 | 110 | 221
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of subjects reporting any AEs
Time Frame: 40 weeks
Population: Safety population: Group 1 and Group 2 consisted of subsets of subjects who received masked treatment with OTX-101 0.09% or with Vehicle, respectively, in OTX-101-2016-001. All subjects received open-label treatment with OTX-101 0.09% in OTX-101-2016-002.
Measure: Number; unit: Count of participants
Groups:
- Group 1; Group 2: OTX-101 0.09%: 0.09% cyclosporine nanomicellar solution
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 129 | 129
Count of participants | 68 | 81

ADVERSE EVENTS:
Time Frame: Day 448
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/129
Serious Adverse Events (participants affected / at risk) | 4/129 | 4/129
Other Adverse Events (participants affected / at risk) | 55/129 | 69/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=129) | Group 2 (N=129)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=129) | Group 2 (N=129)
Conjunctival hyperaemia (Eye disorders) | 12 | 14
Vitreous detachment (Eye disorders) | 5 | 2
Posterior capsule opacification (Eye disorders) | 5 | 1
Blepharitis (Eye disorders) | 3 | 4
Punctate keratitis (Eye disorders) | 12 | 4
Instillation site reaction (General disorders) | 1 | 3
Instillation site lacrimation (General disorders) | 1 | 3
Instillation site pruritus (General disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Eye irritation (Eye disorders) | 2 | 2
Conjunctival haemorrhage (Eye disorders) | 2 | 2
Instillation site pain (General disorders) | 17 | 42
Intraocular pressure increased (Investigations) | 2 | 1
Cataract (Eye disorders) | 2 | 0
Cataract nuclear (Eye disorders) | 2 | 0
Eye allergy (Eye disorders) | 2 | 0
Retinal haemorrhage (Eye disorders) | 2 | 0
Visual acuity reduced (Eye disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT02845674/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02845674/SAP_001.pdf